CLINICAL TRIAL: NCT06689137
Title: Evaluation of the Effect of Dexmedetomidine Infusion on Postoperative Neurocognitive Disorder in Patients Undergoing Laparotomic Abdominal Surgery
Brief Title: Effects of Dexmedetomidine on Postoperative Neurocognitive Disorder
Status: Active, not recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Munevver Duzgun, Specialist Doctor, Anesthesiologist, Haseki Training and Research Hospital
Other Study IDs: HEA-AAR-MK-02
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Neurocognitive Disorder; Dexmedetomidine Infusion; Postoperative Cognitive Dysfunction; Postoperative Cognitive Dysfunction(POCD); Laparoscopic Abdominal Surgery
Keywords: postoperative cognitive dysfunction; peroperative dexmedetomidine infusion; neurocognitive disorder
MeSH Terms: conditions — Neurocognitive Disorders; Postoperative Cognitive Complications | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with dexmedetomidine group: In this study, neurological evaluation tests will be performed before and after surgery for patients who will undergo laparotomic lower and upper gastrointestinal system surgery. All patients will be followed during the perioperative period according to the standards specified in the American Society of Anesthesia guideline. Neurological evaluations will be performed at the 24th hour before surgery, on the day of surgery, and on the 1st, 3rd and 5th days after surgery. Those who underwent total intravenous anesthesia after peroperative anesthesia management will constitute this group. The total amounts of dexmedetomidine, remifentanyl consumed in this group will be recorded.
  Interventions: Other: mini mental state assessment test; Other: mini-cog test
- without dexmedetomidine group: In this study, pre- and postoperative neurological evaluation tests will be performed on patients who will undergo laparotomic lower and upper gastrointestinal system surgery. All patients will be monitored during the perioperative period according to the standards specified in the American Society of Anesthesiologists guide. Neurological evaluations will be performed 24 hours before surgery, on the day of surgery, and on the 1st, 3rd and 5th days after surgery. Those who did not receive dexmedetomidine infusion during peroperative anesthesia management will constitute this group. The total amounts of and remifentanyl consumed in this group will be recorded.
  Interventions: Other: mini mental state assessment test; Other: mini-cog test

INTERVENTIONS:
Other: mini mental state assessment test — Anesthesia management during surgery for this disease in the postoperative period should be carefully planned. It will be important to examine the neurocognitive effects of anesthesia management in the postoperative period in this patient group. In this study, the frequently used Mini mental state assessment test and Mini-cog test will be used. With mini mental state assessment, the patient is asked a number of simple questions to evaluate cognitive functions and each question has certain points. Changes in these score levels preoperatively and postoperatively will be compared within each patient. At the end of the study, preoperative and postoperative changes will be compared statistically between the groups.
  Other Names: neurocognitive disorder assessment
Other: mini-cog test — Anesthesia management during surgery for this disease in the postoperative period should be carefully planned. It will be important to examine the neurocognitive effects of anesthesia management in the postoperative period in this patient group. In this study, the frequently used Mini mental state assessment test and Mini-cog test will be used.With Mini-cog test, the patient is asked a number of simple questions to evaluate cognitive functions and each question has certain points. Changes in these score levels preoperatively and postoperatively will be compared within each patient. At the end of the study, preoperative and postoperative changes will be compared statistically between the groups.
  Other Names: neurocognitive disorder assessment

SUMMARY:
This prospective study involves assessing neurocognitive function in patients undergoing laparotomic gastrointestinal surgery. Mini Mental state Assessment test and Mini-Cog tests will be conducted at multiple intervals preoperatively and postoperatively. Anesthesia management, vital signs, drug consumption, and blood gas values will be recorded throughout the surgery. After all neurocognitive evaluations of the patients are performed at planned intervals for 1 week, the levels of dexmedetomidine and remifentanyl consumed by the patients in the peroperative period will be determined from the anesthesia follow-up sheet and the total duration and amount used will be recorded. At the end of the study, the relationship between neurocognitive values and dexmedetomidine will be compared.

DETAILED DESCRIPTION:
All results of laparotomic gastrointestinal surgery that meet the inclusion criteria of the preoperative anesthesia evaluation process will be determined, and the neurocognitive evaluations, mini mental state assessment test and Mini-cog test will be delivered to all these patients by the anesthesiologist doctor 24 hours before the preoperative period. These two tests will be repeated by the same doctor in the preoperative waiting room on the day of the operation.

From the preoperative waiting room, patients will be taken to the operation room after premedication with 2mg midazolam. After patients are monitored with standard American Society of Anesthesia monitoring (Heart rate (HR), peripheral saturation, non-invasive artery pressure monitoring), patient state index(PSI), the first values will be recorded before surgery. During induction, 1-2mg/kg propofol, 2mcg/kg Fentanyl and 0.8mg/kg rocuronium will be administered and then the patient will be intubated. Patients will be monitored to be normothermic by body temperature monitoring, and Sevoflurane anesthesia will be maintained at 1 Minimal alveolar concentration level as inhalation anesthesia. Patient state index value will be kept between 40-60%. During the peroperative period, non-invasive arterial pressure values, saturation values, heart rate, body temperature values will be recorded on the follow-up form as preoperative, at the beginning of the operation, at 30-minute intervals from the beginning of the operation, and before and after extubation at the end of the operation. If the anesthesiologist starts remifentanyl and dexmedetomidine infusion to the patients during the surgery, when it started and at what dose will be noted on the anesthesia chart. The anesthesiologist performing the neurocognitive evaluation will not be aware of this. The decision whether to start these medications will depend on the relevant anesthesiologist's decision regarding the patient's specific anesthesia management, regardless of the study.

Heart rate, peripheral saturation, non-invasive artery pressure values will be recorded upon entering and exiting the postoperative recovery unit. The patients' total bleeding amount, amount and type of intravenous fluid administered, and blood gas values will be recorded throughout the surgery.

Postoperative pain monitoring will be done with the Numerical Pain Rating Scale, and in patients with an Numerical pain rating scale score greater than 4, Tramadol will be given 100mg every 6 hours, Nonsteroidal anti-inflammatory 100mg every 8 hours, and paracetamol 1000mg every 6 hours will be given intravenously if necessary.

Mini mental state assessment test and Mini-cog test will be repeated in all patients by the anesthesiologist just before being transferred from the postoperative recovery unit to the ward and at the 24th hour, 3rd day, and 5th postoperative day.

After all neurocognitive evaluations of the patients are performed at planned intervals for 1 week, the levels of dexmedetomidine and remifentanyl consumed by the patients in the peroperative period will be determined from the anesthesia follow-up sheet and the total duration and amount used will be recorded.

Anesthesia management of patients during the preoperative and peroperative periods will be planned and implemented as deemed appropriate by the anesthesiologist who follows the patient during the surgical period, regardless of this planned study. The researcher performing the neurocognitive evaluation will not have any intervention or knowledge in these processes. The reason why this study was planned prospectively is that neurocognitive evaluation will be performed prospectively for 1 week. There is no intervention in the patient's anesthesia management and medications, or in the grouping of patients and their treatment. At the end of the study, the relationship between neurocognitive values and dexmedetomidine will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 who will undergo laparotomic lower and upper gastrointestinal system surgery

Exclusion Criteria:

* American society of anesthesia of 4-5 patients
* Patients without voluntary consent
* Patients with previous surgery or vertebrobasilar insufficiency
* Patients with Carotis stenosis
* Patients with a visual analog scale above 4 in the postoperative recovery unit
* Patients whose cerebral oxygenation decreased by 15% from the beginning in cerebral oximetry monitoring during the perioperative period
* Patients with bleeding that disrupts hemodynamics during follow-up and bleeding greater than 20% of body volume
* Patients with postoperative intensive care unit follow-up
* Patients with a decrease of more than 20% from the baseline systolic value (based on ward monitoring) during follow-up
* Patients with intraoperative ventilation failure, patients with hypercarbia, hypocarbia
* Patients whose Patient State Index value falls below 25, which is sufficient for the depth of anesthesia, during anesthesia induction or maintenance.
* Patients with known neurological, psychiatric, unstable cardiovascular, renal or hepatic system disease
* Patients with Uncontrolled Hypertension
* Patients with greater than 1st degree heart block
* Patients allergic to α2 adrenergic receptor agonist
* Patients who cannot speak and do not know Turkish
* Alcohol and substance addicted patients
* Patients who have used opioids in the last 24 hours
* Patients who developed sepsis during postoperative follow-up
* Patients with a history of recurrent surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo laparotomic lower and upper abdominal surgery will constitute the patient groups of this study. Patients who will be operated on due to early stage gastrointestinal tumor will constitute the study population. Among these patients, those without neurological disorders will be included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Decrease in Mini Mental State Assessment test | Preoperative 24 hours before, in the preoperative operating room, at the 1st postoperative hour, on the 1st, 3rd, 5th postoperative days.
  Patients who will undergo laparotomic lower and upper gastrointestinal system surgery will be given a mini mental state assessment test at the preoperative 24th hour, before and after surgery, and on the 1st, 3rd, and 5th postoperative days. In this test, the patient's neurocognitive status will be evaluated by asking simple questions that investigate their mental characteristics. Each question has a score and the total score indicates the patient's condition. In these patients, this test will be repeated at regular intervals after surgery and postoperatively and the results will be recorded. High scores on this test indicate good neurological stability, whereas falling is associated with poor neurological status. Changed in the value as a result of this test will be investigated.

SECONDARY OUTCOMES:
Decrease in Mini-cog Test | Preoperative 24 hours before, in the preoperative operating room, at the 1st postoperative hour, on the 1st, 3rd, 5th postoperative days.
  Mini-cog test will be applied to undergo laparotomic lower and upper gastrointestinal system surgery at the 24th hour before surgery, before and after surgery, and on the 1st, 3rd and 5th days after surgery. In this test, the patient's neurocognitive status will be evaluated by asking simple questions investigating their mental characterise the 24th hour before surgery, before and after surgery, and on the 1st, 3rd and 5th days after surgery. In this test, the patient's neurocognitive status will be evaluated by asking simple questions investigating their mental characteristics. Each question has a score and the total score indicates the patient's condition. In these patients, this test will be repeated at regular intervals during and after surgery and the results will be recorded. High scores on this test indicate good neurological stability, whereas falling is associated with poor neurological status.Changed in value as a result of this test will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Munevver Kayhan, Medical Doctor, Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tufanogullari B, White PF, Peixoto MP, Kianpour D, Lacour T, Griffin J, Skrivanek G, Macaluso A, Shah M, Provost DA. Dexmedetomidine infusion during laparoscopic bariatric surgery: the effect on recovery outcome variables. Anesth Analg. 2008 Jun;106(6):1741-8. doi: 10.1213/ane.0b013e318172c47c. PMID 18499604
- [Background] Maldonado JR, Wysong A, van der Starre PJ, Block T, Miller C, Reitz BA. Dexmedetomidine and the reduction of postoperative delirium after cardiac surgery. Psychosomatics. 2009 May-Jun;50(3):206-17. doi: 10.1176/appi.psy.50.3.206. PMID 19567759